CLINICAL TRIAL: NCT04541238
Title: Imaging Template for Reporting Anal Fistula
Acronym: ITRAF
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Treviso Regional Hospital (Network)
Responsible Party: Principal Investigator, Ugo Grossi, Colorectal Surgeon, Treviso Regional Hospital
Other Study IDs: ITRAF2020
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Novel template report: The last 100 consecutive and anonymized MRI investigations for primary perianal fistula reported according to standard practice by dedicated radiologists (the last 10 reports from each of 10 international centers) are reviewed blindly and independently by two experienced radiologists (based on case load, years of experience and publications on anal fistula) using a novel template incorporating 8 key descriptors.
  A third independent experienced radiologist will resolve any disagreement and assess the presence of descriptors in the original report compared to the novel template.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Magnetic resonance imaging

SUMMARY:
Magnetic resonance imaging (MRI) is the most used diagnostic tool for pre-operative assessment of anal fistula.

However, there is lack of standardization in reporting this investigation. Moreover, reports may miss a number of key information for surgical planning.

The aim of this study is to assess the effectiveness, reproducibility, and acceptability of a new template for reporting anal fistula, which may favor standardization in clinical practice and inform surgical decision making.

ELIGIBILITY:
Inclusion Criteria:

* Adults with primary anal fistula (cryptoglandular or Crohn-related) undergoing MRI

Exclusion Criteria:

* Active cancer of the anorectum
* Recto-vaginal fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 MRI investigations for anal fistula.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the novel template compared to standard reporting based on the number of key descriptors | 60 days

SECONDARY OUTCOMES:
Inter-rater agreement between two independent experienced radiologists using the novel template | 7 days
Qualitative analysis | 30 days
  The 100 MRI investigations (100 original reports and 100 using the novel template) are sent to 20 experienced surgeons (10 randomly selected reports per surgeon, of which 5 reported conventionally and 5 using the novel template), who will complete a semistructured e-mail interview to collect in-depth information about any barriers and facilitators to implementation of the novel template, and ultimately explore surgical decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Grossi, PhD, Principal Investigator — Treviso Regional Hospital, University of Padua
Locations (1):
- Treviso Regional Hospital, Treviso, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD are available on request
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Sudol-Szopinska I, Santoro GA, Kolodziejczak M, Wiaczek A, Grossi U. Magnetic resonance imaging template to standardize reporting of anal fistulas. Tech Coloproctol. 2021 Mar;25(3):333-337. doi: 10.1007/s10151-020-02384-6. Epub 2021 Jan 5. PMID 33400032